CLINICAL TRIAL: NCT02423954
Title: A Phase Ib/II Study of Nivolumab Plus Chemotherapy in Patients With Advanced Cancer (NivoPlus)
Brief Title: Study of Nivolumab Plus Chemotherapy in Patients With Advanced Cancer (NivoPlus)
Acronym: NivoPlus
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator no longer at site to enroll patients or write up data
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WG2015001
Record Dates: First submitted 2015-04-13; First posted 2015-04-22 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Advanced Cancer; Pancreatic Cancer; Renal Cell Cancer; Non Small Cell Lung Cancer; Colorectal Carcinoma; Endometrial; Uterine
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — temsirolimus; Irinotecan; Capecitabine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Temsirolimus 25 mg every 14 days + nivolumab
  Interventions: Drug: Temsirolimus; Drug: nivolumab
- Arm 2 (Experimental): Irinotecan 150 mg/m2 every 14 days + nivolumab
  Interventions: Drug: Irinotecan; Drug: nivolumab
- Arm 3 (Experimental): Irinotecan + capecitabine + nivolumab irinotecan 175 mg/m2 on day 1 every 14 days + capecitabine 1000 mg PO BID days 1-5 on, days 6-7 off, each 7 day period
  Interventions: Drug: Irinotecan + capecitabine; Drug: nivolumab

INTERVENTIONS:
Drug: Temsirolimus
  Other Names: Torisel
  Arms: Arm 1
Drug: Irinotecan
  Other Names: Camptosar
  Arms: Arm 2
Drug: Irinotecan + capecitabine
  Other Names: Camptosar + Xeloda
  Arms: Arm 3
Drug: nivolumab
  Other Names: Opdivo

SUMMARY:
Determine Phase 2 dose of study drug

DETAILED DESCRIPTION:
Determine the recommended phase 2 dose (RP2D) of chemotherapy in combination with nivolumab in subjects with advanced cancer.

ELIGIBILITY:
Inclusion criteria for Phase Ib and II:

1. Patient at least 18 years old and has definitive histologically or cytologically confirmed metastatic solid tumor.
2. Patient has one or more metastatic tumors measurable by CT scan (or PET/CT, if patient is allergic to CT contrast media). Tumor sites that are considered measureable must not have received prior radiation therapy. For metastatic tumors not measurable by CT and/or PET/CT, there needs to be tumor measuring at least 1cm in one dimension by digital calipers on physical exam.
3. Patients can be enrolled only on one of the treatment arms on this trial.
4. The investigator will select the appropriate treatment arm for the patient with the following requirements: (a) Patients cannot have had prior progression or intolerance on the single agent chemotherapy and then enrolled on an arm with that same single agent chemotherapy plus nivolumab (b) The chemotherapy on the arm selected must be considered standard of care or its components listed in the NCCN guidelines (www.nccn.org) for that cancer type.
5. Have recovered from acute toxicities of prior treatment:

   * > 3 weeks must have elapsed since receiving any investigational agent.
   * > 2 weeks must have elapsed since receiving any radiotherapy, or ≥ 3 weeks or 5 half-lives whichever is shorter for treatment with cytotoxic or biologic agents ( ≥ 6 weeks for mitomycin or nitrosoureas). Chronic treatment with non-investigational gonadotropin-releasing hormone analogs or other hormonal or supportive care is permitted.
6. Patient has adequate biological parameters as demonstrated by the following blood counts at time of screening:
7. Absolute neutrophil count (ANC) > 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 9 g/dL. Subject can be given packed red blood cell transfusion
8. Calculated creatinine clearance > 40 ml/min by Cockroft-Gault equation:

   [CreatClear = Sex * ((140 - Age) / (SerumCreat)) * (Weight / 72); where Sex = 1 for men and 0.85 for women], total bilirubin 1.5 times the upper limit of normal (ULN) range, AST/ALT ≤ 3 times the upper limit of normal (ULN) range.
9. Thyroid stimulating hormone (TSH) within institutional normal limits. If TSH is above the upper limit of normal range, then a free T4 within institutional normal limits is acceptable. If thyroid replacement therapy is initiated then patient may be screened and enrolled once the above criterion is met.
10. Persistent prior systemic therapy non-hematologic AE grade ≤ 2 (except alopecia or correctable electrolyte abnormality with supplementation)
11. Patient has a Karnofsky performance status (KPS) ≥ 70.
12. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier method) for the duration of the study and for 5 months following the last dose of nivolumab and 30 days following the last dose of chemotherapy on this trial on this trial, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial. If a female subject or female partner of a male subject becomes pregnant during this period then patient will be recommended to seek appropriate obstetric care. The study will not be monitoring subjects or female partners of subjects for pregnancy after the last dose of study drug or chemotherapy.

Exclusion Criteria for Phase Ib and II:

1. Active clinically serious infection > CTCAE (version 4.03) Grade 2.
2. Serious non-healing wound, ulcer, or bone fracture.
3. Patient has known brain metastases. Baseline imaging of the brain is required within 28 days prior to randomization.
4. Prior therapy with a mammalian target of rapamycin (mTOR) inhibitor for the RCC subjects, prior therapy with irinotecan or topotecan for NSCLC subjects, and prior therapy with irinotecan for CRC patients.
5. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements.
6. Patient has known active infection with HIV, hepatitis B, or hepatitis C (patients are NOT required to be tested for the presence of such viruses prior to therapy on this protocol).
7. Requiring daily corticosteroid dose ≥ 10 mg prednisone or equivalent per day.
8. Patient has undergone major surgery, other than diagnostic surgery (e.g., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
9. Patient has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the patient's safety or the study data integrity.
10. Patient will be receiving any other anti-cancer therapy during participation in this trial.
11. Prior treatment with nivolumab is not allowed. Prior receipt of other PD-1 inhibitors or PD-L1 inhibitors is allowed.
12. Active or prior documented autoimmune disease requiring systemic treatment within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
The recommended phase 2 dose (RP2D) of chemotherapy in combination with nivolumab in subjects with advanced cancer. | up to 4 weeks
  phase 2 dosing of nivolumab + chemotherapy

SECONDARY OUTCOMES:
Frequency of grade 3 or higher treatment-related adverse events by CTCAE 4.03 | up to 12 months
  Identify adverse Events
Response rate by irRC and response evaluation criteria in solid tumors (RECIST) 1.1 criteria1,2 | 12 weeks
  Identify tumor response
The overall survival (OS) and progression-free survival (PFS) | up to 12 months
  Assess time until death after treatment
Quantify changes in amount of blood proteins and circulating tumor DNA in patients enrolled on this study | up to 12 months
  Assess tumor marker levels

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Waypa, MSN, FNP, Study Director — Western Regional Medical Center; Cynthia Lynch, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Cancer Treatment Center of America @ Western Regional Medical Center, Goodyear, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided